CLINICAL TRIAL: NCT04700462
Title: Optimizing Tailored-feedback Message to Promote Adherence Behavior to Prevent COVID-19 in African Americans
Brief Title: COVID-19 Preventive Behavior in African Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00250644; 3R01AG056587-03S1 (NIH)
Record Dates: First submitted 2021-01-06; First posted 2021-01-07 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-01

CONDITIONS: Covid19; Health Behavior
Keywords: COVID-19; Smartphone App; Preventative Behavior; Self-Management; Health Disparities
MeSH Terms: conditions — COVID-19; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sm-EMA (Experimental): Participants will receive the Self-monitoring ecological momentary assessment behavior change tool.
  Interventions: Behavioral: Sm-EMA

INTERVENTIONS:
Behavioral: Sm-EMA — Self-monitoring ecological momentary assessment behavior change tool to promote adherence to a desired behavior (i.e. COVID-19 preventative behaviors).

SUMMARY:
The Center Disease Control has published a set of guidelines to contain the spread of the virus, since it is known to spread from person-to-person. Given the vaccine and specific antiviral treatment for Coronavirus disease (COVID-19) remain under development and will take months or years to develop, intermittent and sustained preventive behaviors may be needed into 2022 unless effective treatments or vaccines are developed. Thus, effectively implementing preventive behaviors remains a critical step in bringing the pandemic under long-term control. Leveraging the ecological momentary assessment (EMA) method developed in the parent R01 for smartphones, which allows for real-time data collection on individual's behaviors, the investigators propose a prospective single arm and longitudinal study to examine the effectiveness of self-monitoring EMA (SM-EMA) in promoting adherence to COVID-19 preventative behaviors. SM-EMA users will download the smartphone app which includes: (1) instructional videos to provide knowledge of preventative behaviors; (2) self-monitoring of preventative behaviors during intervention and follow-up phases; (3) tailored-feedback messages to encourage preventative behaviors; and (4) mobile-enabled website to provide an interactive learning platform. If proven efficacious, this intervention could be efficiently disseminated to reach the larger public and foster preventive behaviors into self-management as effective strategies for long-term control of the COVID-19 pandemic.

DETAILED DESCRIPTION:
Given the vaccine and specific antiviral treatment for COVID-19 will take months or years to develop and finalize, preventive behaviors remain the most effective strategy thus far and may be needed until 2022 to control the pandemic. African Americans, who have 3-fold higher infection rate and 6-fold higher death rate compared to the white counterparts, are an especially vulnerable population to COVID-19. Immediately initiating a project that promotes and maximizes adherence to preventative behaviors is vital to addressing the ongoing COVID-19 pandemic. The investigators propose a prospective single arm and longitudinal study to examine the effectiveness of SM-EMA in promoting adherence to COVID-19 preventative behaviors. The intervention will include two daily pop-up messages during Week 1 (one in the morning and one in the afternoon), one daily pop-message in Week 2, and two pop-up messages a week in Weeks 3 and 4. The duration for the intervention will be four weeks. The study outcomes will be collected at baseline (pre-intervention, T1), post-(completion of the intervention, T2, primary endpoint), and monthly follow-up for three months (T3-T5). The total study duration will be four months.

ELIGIBILITY:
Inclusion Criteria:

* African American aged 60 or older
* Able to read and write English
* Willing to commit to use the smartphone app with the pop-up messages and then four follow-up surveys (total four months).

Exclusion Criteria:

* No children or others aged 59 years or younger

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Change in Knowledge Test score as assessed by a questionnaire | Pre-intervention, Immediately Post-intervention, 1, 2, and 3 months Post-intervention
  It is a measure of one's knowledge of COVID-19 preventative behaviors, with a score range of 0-18, higher scores indicating better knowledge.
Change in Self-efficacy as assessed by self-efficacy questionnaire | Pre-intervention, Immediately Post-intervention, 1, 2, and 3 months Post-intervention
  It is a measure of one's belief that they will be successful in reaching a behavior goal, with 6-items of questionnaire, with a score of 0-60, higher score indicating higher level of self-efficacy.
Change in preventive Behavior Score | Pre-intervention, Daily during intervention week 1 and bi-weekly during intervention weeks 3-4, Immediately Post-intervention, 1, 2, and 3 months Post-intervention
  It is a measure of one's adherence to COVID-19 preventative behaviors, with a score range 0-18, higher score indicating worsening preventive behaviors.
Change in System Usability Scale (SUS) score | Immediately Post-intervention
  It is used to assess the global view of the participant's assessment about usability of SM-EMA, with a score of 1-7, higher score indicting more useable for the app.
Change in Global Impression of Change as assessed by a questionnaire | Immediately Post-intervention, 1, 2, and 3 months Post-intervention
  It is a single item used to assess the participant's perceived behavior change, with a score of 1-7, higher score indicating better global impression of change.

CONTACTS AND LOCATIONS:
Overall Officials: Chao Hsing Yeh, PhD, Principal Investigator — Johns Hopkins School of Nursing
Locations (1):
- Johns Hopkins School of Nursing, Baltimore, Maryland, United States